# HASTA BİLGİLENDİRİLMİŞ GÖNÜLLÜ OLUR FORMU (BGOF)

| ARASTIRMANIN ADI ( CAL | ISMANIN . | ACIK ADI \ |
|------------------------|-----------|------------|

Retrograd intrarenal cerrahide pozisyon taşsızlığı etkiler mi?: Prospektif randomize kontrollü çalışma

Bir araştırma çalışmasına katılmanız istenmektedir. Katılmak isteyip istemediğinize karar vermeden önce araştırmanın neden yapıldığını bilgilerinizin nasıl kullanılacağının çalışmanın neleri içerdiğini ve olası yararlarını risklerini ve rahatsızlık verebilecek konuları anlamanız önemlidir Lütfen aşağıdaki bilgileri dikkatlice okumak için zaman ayırınız.

## **BU ÇALIŞMAYA KATILMAK ZORUNDA MIYIM?**

Bu çalışmaya gönüllü olmanız durumunda katılımınız sağlanacaktır. Katılmaya karar verirseniz, çalışmadan herhangi bir zamanda ayrılmakta özgürsünüz. Bu durum sizin aldığınız tedavinin standardını etkilemeyecektir.

## ÇALIŞMANIN KONUSU VE AMACI NEDİR?

Retrograd intrarenal cerrahi (RIRC), genellikle 2 cm'den küçük böbrek taşları veya bazı durumlarda daha büyük taşlar için tercih edilir. Özellikle başka yöntemlerin uygun olmadığı hastalarda bu tedavi kullanılabilir. RIRC yöntemi gelişen teknolojiyle birlikte daha etkili hale gelmiş olsa da, hastaların %72,9-88,3'ünde taşların tamamen temizlendiği görülmüştür. Ancak bazen böbrekte küçük taş parçaları kalabilir ve bu da gelecekte yeni taş oluşumu riskini artırabilir. RIRC için standart bir tedavi yöntemi bulunmamaktadır. Cerrahi teknik, cerrahın deneyimine ve tercihine bağlı olarak değişiklik gösterebilir. Genellikle standart bir hasta pozisyonu kullanılsa da, bazı durumlarda farklı pozisyonlar da tercih edilmekte ve bu pozisyonlar da etkili ve güvenlidir. Bu çalışma, farklı hastanelerde yapılacak ve planlı bir araştırmadır. Çalışmaya katılacak hastalara araştırma hakkında bilgi verilecek ve gönüllü olmaları halinde dahil edileceklerdir. Hastalar iki gruba ayrılacaktır. Bir grupta cerrahi standart bir pozisyonda yapılacak, diğer grupta ise hastaya biraz farklı bir pozisyon verilecektir (vücut hafif eğik ve cerrahi taraf yukarıda olacak sekilde).

#### **CALISMA İSLEMLERİ**

Hastalarımıza olağan ameliyat süreci dışında ek bir işlem yapılmayacaktır. Çalışmaya alınacak hastalara operasyon sırasında ameliyat masasında ayak ve opere olacak tarafı yukarıda (t-tilt pozisyonu) tutulacak pozisyon verilecek ve takiplerinizde taşlarınızın ne kadarının düşürüldüğü rutin takiplerde olduğu gibi incelenecektir.

#### BENÍM NE YAPMAM GEREKÍYOR?

Ameliyat olmayı ve çalışmaya katılmayı kabul ettiğiniz takdirde, taburculuk sonrası 1. ayda rutin kontrole gelmeniz beklenmektedir

| ÇALIŞMAYA KATILMAMIN NE GİBİ OLASI YAN ETKİLERİ, RİSKLERİ VE RAHATSIZLIKLARI VARDIR? |
|---|
| Çalışmanın, ameliyat ile ilgili onam vermiş olduğunuz risklere ek bir riski bulunmamaktadır. |
| GEBELİK VE DOĞUM KONTROLÜ |
| Operasyonlarımızda ve takip tetkiklerimizde tomografi gibi radyasyon yayan tetkikleri kullanılacağı için gebelik<br>durumunun veya isteğinin olmaması gerekmektedir. |
| ÇALIŞMAYA KATILMANIN OLASI YARARLARI NELERDİR? |
| Çalışmada operasyon sırasında verilecek pozisyonun ameliyat sonrasında böbreğinizde taş kalmama ihtimalini<br>arttıracağını öngörüyoruz. |
| GÖNÜLLÜ KATILIM |
| Bu çalışmaya gönüllü olmanız durumunda katılımınız sağlanacaktır. |
| ÇALIŞMAYA KATILMAMIN MALİYETİ NEDİR? |
| Çalışmanın ek bir maliyeti yoktur. |

| KİŞİSEL BİLGİLERİM NASIL KULLANILACAK? |
|---|
| Araştırma süresince elde edilen bilgiler size özel bir kod numarası ile kaydedilecektir. Her türlü kişisel bilgi gizli tutulacaktır. Araştırmanın sonuçları yalnızca bilimsel amaçla kullanılacaktır. Araştırma yayınlansa bile kimlik bilgileri verilmeyecektir. Ancak, gerektiğinde araştırmanın izleyicileri, etik kurullar ve resmi makamlar bilgilerinize ulaşabilecektir. Siz de istediğinizde bu bilgilere ulaşabileceksiniz. |
| ARAŞTIRMA SÜRESİNCE 24 SAAT ULAŞILABİLECEK KİŞİLER |
| Dr. Murat Gülşen - Tel: 05062357421, Dr. Cemil Aydın - Tel: +90 532 696 03 78, Dr. Ertuğrul Köse - Tel: +90 531 770 73 51, Dr. Utku Gürel Özcan - Tel: +90 539 318 71 20 |
| ÇALIŞMADAN AYRILMAMI GEREKTİRECEK DURUMLAR |
| Bu araştırmaya katılıma izin vermek tamamen sizin isteğinize bağlıdır. Araştırmada yer alınmasına onay verebilir, katılımı onaylamayabilir ya da herhangi bir aşamada araştırmadan ayrılma kararı verebilirsiniz. Araştırmadan çekilmeyi tercih etmeniz ya da araştırıcı tarafından araştırma dışında bırakılma durumunda da, o ana kadar elde edilmiş olan veriler bilimsel amaçla kullanılabilecektir. |
| YENİ BİLGİLER ÇALIŞMADAKİ ROLÜMÜ NASIL ETKİLEYEBİLİR |
| Yeni bilgiler tarafınıza ivedilikle iletilecektir. |
| Çalışmaya Katılma Onayı Bilgilendirilmiş Gönüllü Olur Formundaki tüm açıklamaları okudum. Bana, yukarıda konusu ve amacı belirtilen araştırma ile ilgili yazılı ve sözlü açıklama aşağıda adı belirtilen hekim tarafından yapıldı. Araştırmaya gönüllü olarak katıldığımı, istediğim zaman gerekçeli veya gerekçesiz olarak araştırmadan ayrılabileceğimi ve kendi isteğime bakılmaksızın araştırmacı tarafından araştırma dışı bırakılabileceğimi biliyorum. Söz konusu araştırmaya, hiçbir baskı ve zorlama olmaksızın kendi rızamla katılmayı kabul ediyorum. saklamam için bu belgenin bir kopyasını çalışma sırasında dikkat edeceğim noktaları da içerecek şekilde bana teslim etmiştir |

| Gönüllünün Adı Soyadı / Tarih / İmzası | |
|------------------------------------------------------|---|
| Açıklamaları Yapan Adı Soyadı / Tarih / İmzası | |
| Olur İşlemine Tanık Olan Adı Soyadı / Tarih / İmzası | |
| Yasal Temsilcinin Adı Soyadı / Tarih / İmzası | 1 |